CLINICAL TRIAL: NCT06047340
Title: Feasibility Study for the Use of Computer Game Technology in the Early Diagnosis of Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Feasibility Study of Game Technology in the Early Diagnosis of Mild Cognitive Impairment and Alzheimer's Disease
Acronym: G:DATA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ascentys Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 321523
Record Dates: First submitted 2023-09-02; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Dementia Alzheimers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Interventional study with three study arms (mild cognitive impairment, mild AD-related dementia, healthy controls).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early AD (Experimental): 10 participants with early AD
  Intervention: Game
  Interventions: Device: G:DATA, dementia screen videogame
- MCI (Experimental): 10 participants with mild cognitive impairment
  Intervention: Game
  Interventions: Device: G:DATA, dementia screen videogame
- Health Control (Active Comparator): 10 healthy control participants
  Intervention: Game
  Interventions: Device: G:DATA, dementia screen videogame

INTERVENTIONS:
Device: G:DATA, dementia screen videogame — A videogame for screening

SUMMARY:
This study will test G:DATA, a simple computer game designed to diagnose Alzheimer's Disease, in three different groups of people, some of whom have Alzheimer's Disease. It will look at whether the results of G:DATA match the results of tests that are used to diagnose people with Alzheimer's Disease now. The Investigators will also ask patients and healthcare staff for participant views on the G:DATA game.

DETAILED DESCRIPTION:
Alzheimer's Disease is a type of dementia that causes progressive deterioration to memory, thinking and behaviour. It is currently thought to affect 50 million people globally, although 75% of those affected are thought to be undiagnosed, with no access to treatment.[2] Diagnosis requires extensive clinical evaluation, involving a range of techniques that are resource-intensive and can only be performed in clinical settings. Research has demonstrated a direct link between carefully designed spatial learning within computer games and the detection of deterioration in specific brain cells first affected by Alzheimer's Disease, overlooked by existing assessment techniques. This research will look at the feasibility of using a computer game diagnostic tool, called G:DATA, in the diagnosis of Alzheimer's Disease. It will do this by providing a clinical benchmark, consolidating the results of gameplay performance against current clinical gold-standard assessments, during a clinical study conducted with two patient groups (patients with Mild Cognitive Impairment (MCI), patients with mild AD-related dementia) and a healthy controls group. Outcomes will include validity data of the game's output in diagnosing Alzheimer's Disease, together with data on the tool's usability, and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 55-79 years
* Willing and able to provide informed consen-

Exclusion Criteria:

* A concurrent diagnosis of epilepsy
* A history of severe visual impairment, e.g. macular degeneration, diabetic reti-nopathy, as determined by the clinical team
* A history of head trauma
* Presence of Sleep Apnoea
* History of alcohol dependence
* History of illicit drug use
* Severe upper limb arthropathy
* The use of cognitive enhancing drugs e.g. cholinesterase inhibitors-

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
In Game Navigation Test Score | 9 months
  In Game Navigational Test Score of each participant in correlation to clinical assessment score. This doesn't use any form of scale and higher scores refer to worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hywel Dda University Health Board, Carmarthen, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants will be assigned a unique study ID and data collected will be labelled with the study ID only. An enrolment log will record participant name, date of birth and hospital or NHS number. No personal identifiable information will be included as part of the research dataset leaving the local site for analysis.
Supporting Information: Study Protocol
Time Frame: start date 01/09/23 end date 31/12/23
  I couldn't select the no ipd sharing option
Access Criteria: no one beyond the study team will be able to access data I couldn't select the no ipd sharing option
URL: http://www.ascentys.co.uk